CLINICAL TRIAL: NCT04092439
Title: The Effects of Watermelon Juice Supplementation on Postprandial Vascular Endothelial Function and Blood Flow During Hyperglycemia: A Pilot Study
Brief Title: The Effects of Watermelon Juice Supplementation on Postprandial Vascular Endothelial Function
Acronym: WMJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Timothy Allerton, PhD, Postdoctoral Fellow, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 2019-024
Record Dates: First submitted 2019-09-15; First posted 2019-09-17 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Endothelial Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Watermelon juice (Experimental): The study participants consumed 500 ml of 100% watermelon juice for two weeks
  Interventions: Dietary Supplement: Watermelon Juice
- Placebo (Placebo Comparator): The study participants consumed a watermelon flavored, fructose matched control
  Interventions: Dietary Supplement: Watermelon Juice

INTERVENTIONS:
Dietary Supplement: Watermelon Juice — 100% Watermelon Juice

SUMMARY:
The purpose of this study is to test if watermelon juice supplementation improves vascular dysfunction experience during hyperglycemia.

DETAILED DESCRIPTION:
The objective of this pilot study is to determine the potential for watermelon juice to attenuate the reduction postprandial endothelial function and skeletal muscle microvascular blood flow (MVBF) experienced during hyperglycemia.

The investigators will attempt to answer the following hypotheses:

Hypothesis 1: Watermelon juice supplementation will attenuate the reduction in endothelial dysfunction and microvascular blood flow during an oral glucose challenge.

Hypothesis 2: Watermelon juice will increase L-arginine bioavailability during hyperglycemia and correlate with improved vascular response.

Exploratory Aim: The postprandial period is defined by increased sympathetic nervous system activity (vasoconstriction) and NO• mediated vasodilation. Heart rate variability (HRV) is a measurement of the balance of parasympathetic to sympathetic activity. The investigators will measure HRV during the oral glucose challenge to interrogate the possibility that watermelon juice can modulate the balance of blood vessel constriction and relaxation during an oral glucose

Procedures Involved

There will be 1 screening visit, and 2 outpatient visits. Participants will consume watermelon juice or placebo for 2 weeks. The washout period will last 2 weeks prior to the cross-over to the opposite condition. Participants visits will be conducted at the Vascular and Resting Metabolism Lab located in the department of kinesiology at LSU.

Screening Visit

Participants will undergo consenting and fasting blood draws to measure glucose, lipids, and CBC. Vital signs (blood pressure, body weight, body composition (DXA), heart rate, etc) will be measured. For DXA procedure participants will undergo a whole body scan lasting approximately 10 minutes. Participants will remove all metal objects from their body and lie down on the table. The legs will be secured together using two Velcro straps. The participant will be instructed to remain completely still during the scan. Randomization will be performed to allocate the study participant for their initial group assignment to either the watermelon juice group or placebo. The initial six participants will be assigned treatment A for phase 1 and treatment B for phase 2, thereafter the following 6 will be assigned treatment B first then treatment A. The remaining participant will be randomly assigned either treatment A or B in a counterbalanced fashion.

Daily Juice Drop-in visits

Since the required supplementation duration is 14 days participants will be provided with 2 days (Saturday and Sunday) worth of watermelon juice or placebo to account for days when the LSU AG Center will not be open. To allow for scheduling conflicts and unforeseen circumstances a 3 day period of supplementation less then or greater than the 14 periods will be permitted. Participants will also be provided with juice or placebo for anticipated instances where they cannot be on campus. In order to monitor compliance participants will be asked return the juice container for the days where juice was consumed off premises.

Visit 2 and 3: Oral Glucose Challenge - Postprandial FMD and MVBF

Participants will arrive in morning at 6:00am fasted for 10-hours. Body composition will be measured by DXA. Next, participants will rest for 30 minutes in the supine positing while wearing a heart rate monitor (Zephyr, Bioharness) to measure heart rate and heart rate variability. Resting metabolic rate will be measured via indirect calorimetry for 20 minutes. Then fasting measures of blood glucose, FMD (ultrasound) and MVBF (near-infrared spectroscopy) will be taken followed by ingestion of 75 g of glucose (glucola). An IV line will be placed in the participants arm vein for blood draw purposes and will remain there throughout the testing. A blood sample will be drawn, and then the participant will drink a sugar solution consisting of 75 grams of glucose. Blood will be drawn at specific times after the participant consumes the drink. Each blood sample will be about 1 tablespoon. (6 tablespoons total for the test). During the IV procedure, a small amount of the participant's own blood (less than 1 teaspoon) will immediately be returned into the participants vein through the IV after each specimen is collected. Blood will be drawn at minute 15, 30, 60, 90, 120 minutes. Postprandial measurements of FMD and MVBF will be taken at 30, 60, 90, and 120 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Capable and willing to give written informed consent and understand inclusion and exclusion criteria.
2. 18-40 years of age
3. BMI between 18-29.9 kg/m2
4. Willing to allow researchers to draw blood and conduct imaging (DXA) for research purposes.

Exclusion Criteria:

1. Evidence or self-reported history of type 1 or 2 diabetes mellitus
2. Self-reported family history of type 2 diabetes (first degree relative with type 2 diabetes)
3. Evidence or self-report history of deep vein thrombosis, pulmonary embolism, cardiovascular, peripheral vascular, cerebral vascular, pulmonary, or renal disease
4. Allergy to watermelon
5. Use of medication known to influence study outcomes, such as:

   1. Insulin
   2. Anti-diabetics (metformin)
   3. Corticosteroids
   4. Beta-blockers
   5. Anti-coagulates
6. Use of supplements known to influence study outcomes, such as;

   1. Beta-alanine
   2. L-arginine
   3. L-citrulline
7. Active smoking

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy D Allerton, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baena-Diez JM, Penafiel J, Subirana I, Ramos R, Elosua R, Marin-Ibanez A, Guembe MJ, Rigo F, Tormo-Diaz MJ, Moreno-Iribas C, Cabre JJ, Segura A, Garcia-Lareo M, Gomez de la Camara A, Lapetra J, Quesada M, Marrugat J, Medrano MJ, Berjon J, Frontera G, Gavrila D, Barricarte A, Basora J, Garcia JM, Pavone NC, Lora-Pablos D, Mayoral E, Franch J, Mata M, Castell C, Frances A, Grau M; FRESCO Investigators. Risk of Cause-Specific Death in Individuals With Diabetes: A Competing Risks Analysis. Diabetes Care. 2016 Nov;39(11):1987-1995. doi: 10.2337/dc16-0614. Epub 2016 Aug 4. PMID 27493134
- [Background] Berrington de Gonzalez A, Hartge P, Cerhan JR, Flint AJ, Hannan L, MacInnis RJ, Moore SC, Tobias GS, Anton-Culver H, Freeman LB, Beeson WL, Clipp SL, English DR, Folsom AR, Freedman DM, Giles G, Hakansson N, Henderson KD, Hoffman-Bolton J, Hoppin JA, Koenig KL, Lee IM, Linet MS, Park Y, Pocobelli G, Schatzkin A, Sesso HD, Weiderpass E, Willcox BJ, Wolk A, Zeleniuch-Jacquotte A, Willett WC, Thun MJ. Body-mass index and mortality among 1.46 million white adults. N Engl J Med. 2010 Dec 2;363(23):2211-9. doi: 10.1056/NEJMoa1000367. PMID 21121834
- [Background] Avogaro A. Postprandial glucose: marker or risk factor? Diabetes Care. 2011 Oct;34(10):2333-5. doi: 10.2337/dc11-1442. No abstract available. PMID 21949226
- [Background] Enkhmaa B, Ozturk Z, Anuurad E, Berglund L. Postprandial lipoproteins and cardiovascular disease risk in diabetes mellitus. Curr Diab Rep. 2010 Feb;10(1):61-9. doi: 10.1007/s11892-009-0088-4. PMID 20425069
- [Background] Keske MA, Premilovac D, Bradley EA, Dwyer RM, Richards SM, Rattigan S. Muscle microvascular blood flow responses in insulin resistance and ageing. J Physiol. 2016 Apr 15;594(8):2223-31. doi: 10.1113/jphysiol.2014.283549. Epub 2015 Jan 12. PMID 25581640
- [Background] Vincent MA, Barrett EJ, Lindner JR, Clark MG, Rattigan S. Inhibiting NOS blocks microvascular recruitment and blunts muscle glucose uptake in response to insulin. Am J Physiol Endocrinol Metab. 2003 Jul;285(1):E123-9. doi: 10.1152/ajpendo.00021.2003. PMID 12791603
- [Background] Williams SB, Cusco JA, Roddy MA, Johnstone MT, Creager MA. Impaired nitric oxide-mediated vasodilation in patients with non-insulin-dependent diabetes mellitus. J Am Coll Cardiol. 1996 Mar 1;27(3):567-74. doi: 10.1016/0735-1097(95)00522-6. PMID 8606266
- [Background] Johnstone MT, Creager SJ, Scales KM, Cusco JA, Lee BK, Creager MA. Impaired endothelium-dependent vasodilation in patients with insulin-dependent diabetes mellitus. Circulation. 1993 Dec;88(6):2510-6. doi: 10.1161/01.cir.88.6.2510. PMID 8080489
- [Background] Tessari P, Cecchet D, Cosma A, Vettore M, Coracina A, Millioni R, Iori E, Puricelli L, Avogaro A, Vedovato M. Nitric oxide synthesis is reduced in subjects with type 2 diabetes and nephropathy. Diabetes. 2010 Sep;59(9):2152-9. doi: 10.2337/db09-1772. Epub 2010 May 18. PMID 20484137
- [Background] Forstermann U. Janus-faced role of endothelial NO synthase in vascular disease: uncoupling of oxygen reduction from NO synthesis and its pharmacological reversal. Biol Chem. 2006 Dec;387(12):1521-33. doi: 10.1515/BC.2006.190. PMID 17132097
- [Background] Deveaux A, Pham I, West SG, Andre E, Lantoine-Adam F, Bunouf P, Sadi S, Hermier D, Mathe V, Fouillet H, Huneau JF, Benamouzig R, Mariotti F. l-Arginine Supplementation Alleviates Postprandial Endothelial Dysfunction When Baseline Fasting Plasma Arginine Concentration Is Low: A Randomized Controlled Trial in Healthy Overweight Adults with Cardiometabolic Risk Factors. J Nutr. 2016 Jul;146(7):1330-40. doi: 10.3945/jn.115.227959. Epub 2016 Jun 8. PMID 27281800
- [Background] Schulman SP, Becker LC, Kass DA, Champion HC, Terrin ML, Forman S, Ernst KV, Kelemen MD, Townsend SN, Capriotti A, Hare JM, Gerstenblith G. L-arginine therapy in acute myocardial infarction: the Vascular Interaction With Age in Myocardial Infarction (VINTAGE MI) randomized clinical trial. JAMA. 2006 Jan 4;295(1):58-64. doi: 10.1001/jama.295.1.58. PMID 16391217
- [Background] Agarwal U, Didelija IC, Yuan Y, Wang X, Marini JC. Supplemental Citrulline Is More Efficient Than Arginine in Increasing Systemic Arginine Availability in Mice. J Nutr. 2017 Apr;147(4):596-602. doi: 10.3945/jn.116.240382. Epub 2017 Feb 8. PMID 28179487

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Watermelon Juice Drink, Then Placebo: Participants first received 500 ml of watermelon juice for the first 2 weeks. After a 2 week washout, they then received 500 ml of a watermelon-flavored placebo drink.
- Experimental: Placebo, Then Watermelon Juice Drink: Participants first received 500 ml of watermelon flavor placebo drink for two weeks. After a 2 week washout, participants then received 2 week of 500 ml of watermelon juice for daily consumption.
Period: Overall Study
Arm/Group | Experimental: Watermelon Juice Drink, Then Placebo | Experimental: Placebo, Then Watermelon Juice Drink
Started | 10 | 8
Completed | 10 | 7
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: The study participants were young and healthy adults with no medical conditions.
Groups:
- Watermelon Juice First, Then Placebo: 100% watermelon juice
  Watermelon Juice: 100% Watermelon Juice
- Placebo First Then, Watermelon Juice: Fructose matched control
  Watermelon Juice: 100% Watermelon Juice
- Total: Total of all reporting groups
Arm/Group | Watermelon Juice First, Then Placebo | Placebo First Then, Watermelon Juice | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.4 (2.7) | 24.2 (3.4) | 23.8 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 2 | 4 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 8 | 18
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 21.9 (1.6) | 25.0 (3.9) | 23.3 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Function
Description: Flow mediated dilation
Time Frame: Two weeks
Population: Young healthy adults
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Placebo: 500 ml of watermelon flavored drink
- Watermelon Juice: Young healthy adults
Arm/Group | Placebo | Watermelon Juice
Number analyzed (Participants) | 17 | 17
millimeters | 3.31 (0.65) | 3.53 (.65)

2. Secondary Outcome: Postprandial Blood Flow
Description: microvascular blood flow
Time Frame: Two weeks
Population: Young healthy adults
Measure: Mean (Standard Deviation); unit: 100 ml tissue/min
Arm/Group | Placebo | Watermelon Juice
Number analyzed (Participants) | 17 | 17
100 ml tissue/min | 36.0 (20.5) | 51.0 (29.1)

ADVERSE EVENTS:
Time Frame: Two weeks for each intervention.
Description: All participants undergoing the intervention were monitored to adverse events.
Groups:
- Placebo: Fructose matched control
  Watermelon Juice: 100% Watermelon Juice
Arm/Group | Watermelon Juice | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT04092439/Prot_000.pdf
  • Informed Consent Form (2019-05-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT04092439/ICF_001.pdf